CLINICAL TRIAL: NCT01434719
Title: Spatial and Temporal Associations Between Human Streptococcus Suis Infections and Pig Diseases in Northern Vietnam, 2010
Brief Title: Human Suis and Pig Diseases in Northern Vietnam
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Responsible Party: Sponsor
Other Study IDs: 02ZN
Record Dates: First submitted 2011-04-06; First posted 2011-09-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Streptococcus Suis Infection
Keywords: Streptococcus suis; Sepsis; Porcine Respiratory and Reproductive System virus; Pig disease; Epidemiology
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- S.suis cases: This group consists of human cases with S.suis infection (confirmed or probable) admitted to National Hospital for Tropical Diseases in 2010.
- Sepsis controls: This group consists of hospital controls diagnosed with sepsis (not caused by S.suis) admitted to National Hospital for Tropical Diseases in 2010.

SUMMARY:
This study aim to test the hypothesis that human S.suis infections are associated in time and space with outbreaks of Porcine Reproductive and Respiratory Syndrome (PRRS) virus or other diseases in pigs.

DETAILED DESCRIPTION:
Streptococcus suis is a zoonotic agent which can cause severe systemic infection in humans exposed to infected pigs or pig derived products. Over 700 cases have been reported worldwide, most of them were in China and Vietnam in the last few years.

In Vietnam, S. suis infection in adults is common, and patients with S.suis are often admitted to the National Hospital for Tropical Diseases (NHTD), a tertiary referral hospital for infectious diseases in northern Vietnam. In 2007, 50 laboratory confirmed cases with S.suis were reported at this hospital, and in 2010, 65 laboratory confirmed S.suis cases have been identified by September. Pig breeding and pork consumption is popular in Vietnam, with the majority of pigs and meat supply channelled from small-scaled un-controlled farmers and slaughterhouses, which pose a great potential health risk to people involved in the chain. A case-control study conducted in southern Vietnam showed that occupational exposure, raising pigs at home and consuming high-risk dishes from pigs significantly increased the risk of S. suis infection.

It has been suggested that the incidence of human S. suis cases is possibly linked to the occurrence of Porcine Respiratory and Reproductive System (PRRS) virus outbreaks in northern Vietnam. In 2010, the disease has spread to over 30 provinces over the country, with many outbreaks reported in northern provinces in the period from April to July. Field observations in other countries showed that PRRS virus infection increased pig's susceptibility to S. suis infection, including serotype 2 and 7. Therefore, PRRS virus outbreaks might have increased the risk of S. suis transmission to humans through exposure to pigs with PRRS virus infection and concomitant S. suis disease. Nevertheless, sufficient data are not available to confirm or refute this hypothesis. Knowledge of spatial and temporal relationships between human S.suis infections and disease outbreaks in pigs can increase our understanding of risk factors for human S.suis infection and support disease prevention and preparedness in the community.

ELIGIBILITY:
Group 1: cases

Inclusion Criteria:

* Date of specimen (blood or CSF sample) collection is between 01/01/2010 to 31/12/2010; and
* S.suis infection confirmed by either CSF or blood culture or PCR; or
* Meet the criteria for a probable case as above (in absence of laboratory confirmation).

Exclusion Criteria:

- Unable to collect patient's spatial data at commune level.

Group 2: controls

Inclusion Criteria:

* Diagnosis as sepsis at hospital admission (based on clinical symptoms or laboratory evidence)
* Admission date between 01/01/2010 and 31/12/2010

Exclusion Criteria:

* Symptoms of meningitis
* Clinically a high suspicion of S. suis infection (culture and PCR negative) as determined by doctor.
* Laboratory culture or PCR result positive for S.suis infection
* HIV infection
* Unable to collect patient's spatial data at commune level

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population under study is the population from which cases of S.suis infection admitted to NHTD arise. Sepsis patients are selected to present the population of interest under the following assumptions:
  * they are representative of the background exposure rate of the population from which cases come from,
  * their diagnosis is independent of the exposure of interest,
  * they are similar to the S.suis cases in terms of care seeking and referral patterns.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Temporal proximity to the nearest pig outbreak of human cases versus human controls | Up to 1 year
  The number of days separating identified nearest pig outbreak and identified human cases of S. suis versus the number of days separating identified nearest pig outbreak and human controls.
Spatial proximity to the nearest pig outbreak of human cases versus human controls | Up to 1 year
  The number of kilometers separating the identified nearest pig outbreak and identified human cases of S. suis versus the number of kilometers separating the identified nearest pig outbreak and human controls.

SECONDARY OUTCOMES:
Number of human S. suis cases | One year
  Total number of human S.suis cases recorded at NHTD in 2010.
Number of pig disease outbreaks | One year
  Total number of pig outbreaks identified within 2010 in the Northern region.

CONTACTS AND LOCATIONS:
Overall Officials: Kinh V Nguyen, PhD, Principal Investigator — National Hospital for Tropical Diseases; Heiman F Wertheim, PhD, Principal Investigator — Oxford University Clinical Research Unit - Hanoi
Locations (1):
- National Hospital for Tropical Diseases, Hanoi, Hanoi, Vietnam

REFERENCES:
- See also: OUCRU studies public site — http://www.oucru.org/index.php?option=com_content&view=article&id=337&std=02ZN&ox=&cd=02ZN&type=&fil=&inv=&en=&vn=&ran=0.6927202849331444